CLINICAL TRIAL: NCT03479944
Title: Clinical Evaluation of FLACS (Femtosecond Laser Assisted Cataract Surgery) With Combination of LenSx® and Centurion®
Brief Title: Clinical Evaluation of FLACS With Combination of LenSx® and Centurion®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTB258-P001
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FLACS (Experimental): Femtosecond laser assisted cataract surgery (FLACS) in 1 eye, with manual conventional surgery in the fellow eye, as randomized
  Interventions: Procedure: FLACS; Device: CENTURION® Vision System; Device: LenSx®
- Conventional (Active Comparator): Manual conventional surgery in 1 eye, with FLACS in the fellow eye, as randomized
  Interventions: Procedure: Manual conventional surgery; Device: CENTURION® Vision System

INTERVENTIONS:
Procedure: FLACS — Femtosecond laser assisted cataract surgery consisting of LenSx® and Centurion® combination
  Arms: FLACS
Procedure: Manual conventional surgery — Removal of cataractous lens by phacoemulsification
  Arms: Conventional
Device: CENTURION® Vision System — Phacoemulsification aspiration platform for use during cataract surgery
Device: LenSx® — Femtosecond laser system used for continuous curvilinear capsulorhexis (CCC) and lens fragmentation during cataract surgery
  Arms: FLACS

SUMMARY:
The purpose of this study is to evaluate cumulative dissipated energy (CDE), endothelial cell loss, and average torsional amplitude with combination of LenSx® and Centurion® compared to conventional cataract surgery.

DETAILED DESCRIPTION:
Subjects will attend 7 scheduled visits: 1 pre-operative, 1 operative, and 5 post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Cataracts (Grade 2-4 of Emery-Little Classification) with planned cataract removal by phacoemulsification in both eyes;
* Able to comprehend and willing to sign informed consent and complete all required postoperative follow-up procedures;
* Calculated lens power within the available range;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any pathology that could reduce visual potential;
* Hypotony or the presence of a corneal implant;
* Residual, recurrent, active ocular or eyelid disease;
* Poorly dilating pupil;
* Any contraindication to cataract;
* Eyes with two different levels of cataract grade;
* Pregnant, or planned pregnancy during the study;
* Expected to require an ocular surgical treatment at any time during the study;
* Other protocol-specified exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division
Locations (1):
- Alcon Investigative Site, Iizuka, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 57 enrolled subjects, 2 subjects discontinued the study before surgery on the first operated eye. This reporting group includes all subjects for which cataract surgery was performed with the test device (regardless of success or failure) (Treatment-Emergent Safety Analysis Set)
Units Other Than Participants: eyes
Groups:
- All Study Subjects: Cataract extraction surgery with either FLACS or conventional technique allocated to each eye (within-subject), as randomized. Both eye surgeries occurred on the same day.
Period: Overall Study
Arm/Group | All Study Subjects
Started | 55; 110 eyes
FLACS (left or right eye) | 55; 55 eyes
Conventional (fellow eye) | 55; 55 eyes
Full Analysis Set | 53; 106 eyes
Completed | 55; 110 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Treatment Emergent Safety Analysis Set
Arm/Group | All Study Subjects
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (6.6)
Age, Customized [Number; unit: years]
  Less than 60 | 0
  60-69 | 15
  70-79 | 30
  80 and greater | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 55

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Dissipated Energy (CDE)
Description: CDE is not expressed in standard units such as Watts or Joules and accounts for the power and time of longitudinal and torsional ultrasound delivery modes. CDE (the sum total of phacoemulsification energy dissipated at the incision point during the removal of cataractous lens with Centurion® Vision System footpedal in Position 3) was calculated by the Centurion® Vision System as follows: CDE = (Longitudinal time) x (Average longitudinal power) + (Torsional time x 0.4 x Average torsional amplitude). A lower CDE value indicates that less energy was expended in the eye.
Time Frame: Day 0 (operative day)
Population: All eyes with successful cataract surgery for which anterior capsulotomy and lens fragmentation have been completed using the assigned surgical techniques (Full Analysis Set).
Measure: Mean (Standard Deviation); unit: unitless
Units Other Than Participants: eyes
Groups:
- FLACS: Femtosecond laser assisted cataract surgery (FLACS) with LenSx® and Centurion® Vision System in combination
- Conventional: Manual cataract surgery with Centurion® Vision System
Arm/Group | FLACS | Conventional
Number analyzed (Participants) | 53 | 53
Number analyzed (eyes) | 53 | 53
unitless | 0.213 (0.334) | 1.718 (0.898)
Statistical Analysis 1: Comparison: FLACS vs Conventional; Test type: Superiority; p < 0.0001, t-test based on MMRM; MMRM: Mixed Model for Repeated Measures; Least Squares Mean Difference = -1.505, 95% CI 2-sided [-1.720 to -1.289] — Least Squares Mean Difference from a Mixed Model for Repeated Measures

2. Secondary Outcome: Percent Change of Corneal Endothelial Cell Density (ECD) at Visit 5 (150-210 Days After Surgery) From Pre-Operative Visit
Description: Central endothelial cell counts were assessed using specular microscopy. ECD was measured in cells per square millimeter (mm2). The endothelium maintains corneal hydration, and positive percent change value indicates an improvement. In turn, a less negative percent change value is preferable over a more negative percent change value.
Time Frame: Preoperative, Day 150-210 (post-operative)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: eyes
Groups:
- FLACS: Femtosecond laser assisted cataract surgery with LenSx® and Centurion® Vision System in combination
Arm/Group | FLACS | Conventional
Number analyzed (Participants) | 53 | 53
Number analyzed (eyes) | 53 | 53
percent change | -1.5 (5.6) | -2.7 (5.2)
Statistical Analysis 1: Comparison: FLACS vs Conventional; Test type: Superiority; p = 0.2602, t-test based on MMRM; MMRM: Mixed Model for Repeated Measures; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.9 to 3.3] — Least Squares Mean Difference from a Mixed Model for Repeated Measures

3. Secondary Outcome: Percentage of Average Torsional Amplitude
Description: Torsional amplitude (the amplitude of the oscillations of the phacoemulsification tip) was reported on the Centurion® Vision System interface as a percentage from 0 to 100, where 100 represents maximum amplitude. A lower percentage value indicates greater efficiency in the phacoemulsification process.
Time Frame: Day 0 (operative day)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of avg torsional amplitude
Units Other Than Participants: eyes
Arm/Group | FLACS | Conventional
Number analyzed (Participants) | 53 | 53
Number analyzed (eyes) | 53 | 53
percentage of avg torsional amplitude | 19.57 (16.02) | 31.09 (6.56)
Statistical Analysis 1: Comparison: FLACS vs Conventional; Test type: Superiority; Least Squares Mean Difference = -11.52, 95% CI 2-sided [-15.87 to -7.18] — Least Squares Mean Difference from a Mixed Model for Repeated Measures

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of initial treatment through study conclusion, for an average individual duration of 150 to 120 days.
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (test article).
Groups:
- Ocular Adverse Events - FLACS: All subjects/eyes for which cataract surgery was performed with FLACS (regardless of success or failure)
- Ocular Adverse Events - Conventional: All subjects/eyes for which cataract surgery was performed with Conventional technique (regardless of success or failure)
- Non-Ocular Adverse Events: All subjects for which cataract surgery was performed (regardless of success or failure)
Arm/Group | Ocular Adverse Events - FLACS | Ocular Adverse Events - Conventional | Non-Ocular Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 2/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ocular Adverse Events - FLACS (N=55) | Ocular Adverse Events - Conventional (N=55) | Non-Ocular Adverse Events (N=55)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | NA | 1
Epilepsy (Nervous system disorders) | 0 | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03479944/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT03479944/SAP_001.pdf